CLINICAL TRIAL: NCT04098510
Title: Concentration of Mitoquinone Mesylate in Skeletal Muscle After a Single Oral Dose of MitoQ
Brief Title: Concentration of MitoQ in Human Skeletal Muscle
Acronym: MitoQ/muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MitoQ
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Mitochondria-targeted antioxidant; Skeletal muscle biopsies
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MitoQ (Experimental): Subjects ingest 160 mg of MitoQ
  Interventions: Dietary Supplement: MitoQ

INTERVENTIONS:
Dietary Supplement: MitoQ — Subjects ingest 8x20 mg MitoQ capsules

SUMMARY:
The purpose of this study is to determine mitoquinone mesylate concentration levels in skeletal muscle samples obtained after intake of an acute oral dose of MitoQ.

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* Male
* 18-40 years of age

Exclusion Criteria:

* Previous use of MitoQ or CoQ-10 within 30 days of screening appointment
* Ongoing use of MitoQ
* Smoking
* Ongoing treatment with medications
* Disease deemed by the MD to infer a risk to participate in the trial

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Muscle mitoquinone mesylate concentration | Before oral administration of MitoQ
  Concentration of mitoquinone mesylate in skeletal muscle
Muscle mitoquinone mesylate concentration | 1 hours after oral administration of MitoQ
  Concentration of mitoquinone mesylate in skeletal muscle
Muscle mitoquinone mesylate concentration | 3 hours after oral administration of MitoQ
  Concentration of mitoquinone mesylate in skeletal muscle
Muscle mitoquinone mesylate concentration | 5 hours after oral administration of MitoQ
  Concentration of mitoquinone mesylate in skeletal muscle

SECONDARY OUTCOMES:
Blood mitoquinone mesylate concentration | Before as well as 0.5, 1, 1.5, 2, 3, 4 and 5 hours after oral administration of MitoQ
  Concentration of mitoquinone mesylate in venous blood

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No